CLINICAL TRIAL: NCT01311700
Title: Effect of METOprolol in CARDioproteCtioN During an Acute Myocardial InfarCtion. The ME"Effect of METOprolol in CARDioproteCtioN During an Acute Myocardial InfarCtion" (METOCARD-CNIC): A Randomized, Controlled Parallel-group, Observer-blinded Clinical Trial of Early Pre-reperfusion Metoprolol Administration in ST-segment Elevation Myocardial infarctionTOCARD-CNIC Trial.
Brief Title: Effect of METOprolol in CARDioproteCtioN During an Acute Myocardial InfarCtion. The METOCARD-CNIC Trial.
Acronym: METOCARD-CNIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government); Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METOCARD-CNIC; CNIC translational Grant 2009 (Other Grant/Funding Number: CNIC translational Grant 2009 (Exp# 01-2009)); 2010-019939-35 (EudraCT Number); Ministerio de Sanidad (Other Grant/Funding Number: Ministerio de Sanidad, Política Social e Igualdad Grant (EC10-042).)
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2017-12

CONDITIONS: Myocardial Infarction
Keywords: Ischemia; Reperfusion; Myocardial infarction; Beta blockers; Metoprolol; Acute myocardial infarction; Necrosis; Salvaged Myocardium
MeSH Terms: conditions — Myocardial Infarction; Ischemia; Necrosis | interventions — Injections; Metoprolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early metoprolol initiation strategy (Active Comparator)
  Interventions: Drug: Injectable (i.v.) metoprolol tartrate (up to 15 mg).
- Delayed metoprolol initiation strategy (No Intervention)

INTERVENTIONS:
Drug: Injectable (i.v.) metoprolol tartrate (up to 15 mg). — Patients are randomized to active intervention (early metoprolol initiation strategy) or no treatment (delayed metoprolol initiation strategy).
  Patients randomized to early metoprolol initiation strategy receive up to three 5mg i.v. dosages (2 minutes apart) before reperfusion.
  Patients randomized to delayed metoprolol initiation strategy receive no active treatment before reperfusion.
  Patients in both groups receive oral metoprolol tartrate treatment (25-100mg/12h), starting 12-24 hr post-reperfusion.
  Arms: Early metoprolol initiation strategy

SUMMARY:
The purpose of this study is to test whether early pre-reperfusion metoprolol administration in patients suffering and acute myocardial infarction might reduce the size of myocardial necrosis.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a chief cause of death worldwide. The best strategy to limit myocardial damage is to perform an early coronary reperfusion. However, despite reperfusion, the size of infarctions is many times large. Infarct size has been recently shown to be a strong predictor of future cardiovascular events and mortality. Therefore interventions aimed at reducing infarct size are the matter of intense research; but despite great efforts, no therapy has been shown to consistently limit infarct size.

ß-blockers are a class of drugs that have been used to treat cardiovascular conditions for several decades. β-blockers reduce mortality when administered after an AMI, and are a class IA indication in this context. What remains unclear is what timing and route of β-blocker administration gives the maximum cardioprotective effect. In particular, whether early β-blocker administration is able to reduce infarct size is a subject of debate. Recent experimental data suggest that the β1 selective blocker metoprolol is able to limit the area of necrosis only when administered before reperfusion.

The objective of this trial is to determine whether the administration of intravenous pre-reperfusion metoprolol might reduce infarct size.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed* acute anterior wall myocardial infarction (ST segment elevation ≥ 2mm in ≥ 2 contiguous leads [one of which should be V2, V3, or V4]).
2. Killip class I or II on diagnosis.

   * Cases of non-confirmed infarction by enzymatic release (above 2 standard deviations from upper limit of CK and Troponin) are excluded from efficacy analysis but kept in the safety analysis.

Exclusion Criteria:

1. COPD or asthma on active bronchodilator therapy
2. Active treatment with beta blockers
3. Left bundle branch block or pacemaker.
4. Systolic blood pressure <120 mmHg, Heart rate <60 bpm, or AV block (PR˃240 mS or superior) on diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Infarct size evaluated primarily by area of delayed enhancement on cardiac magnetic resonance imaging. | 5-7 days after reperfusion

SECONDARY OUTCOMES:
Infarct size evaluated primarily by the area under the curve of CK, CK-MB and troponin release over the first 72 hours of reperfusion. | over the first 72 hours of reperfusion.
Infarct size evaluated by area of delayed enhancement on cardiac magnetic resonance imaging. | at month 6
Infarct size evaluated by area of delayed enhancement on cardiac magnetic resonance imaging in patients with coronary TIMI flow 0-1 of culprit coronary artery. | 5-7 days after reperfusion.
Percent salvaged myocardium evaluated by cardiac magnetic resonance imaging. | 5-7 days after reperfusion
Recovery of myocardial contraction assessed by magnetic resonance imaging and echocardiography. | at month 6
Myocardial perfusion evaluated by magnetic resonance imaging. | 5-7 days post-reperfusion.
Composite of death, malignant ventricular arrhythmias, reinfarction or admission due to heart failure | hospital discharge, 1, 6 and 12 months post-reperfusion.
Major cardiovascular events (death, malignant ventricular arrhythmias, AV block, cardiogenic shock, reinfarction). | within first 24 hr post-reperfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Borja Ibanez, MD PhD, Principal Investigator — CNIC
Locations (12):
- Spain (12):
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de Vigo-Hospital Meixoeiro, Vigo, Pontevedra
  - Servicio de Urgencias Sanitarias 061 de Galicia, Vigo, Pontevedra
  - Hospital de León, León
  - Hospital La Princesa, Madrid
  - Servicio de Asistencia Municipal de Urgencia y Rescate (SAMUR), Madrid
  - • Centro Nacional de Investigaciones Cardiovasculares Carlos III (CNIC),, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Servicio de Urgencia Médica de la Comunidad de Madrid (SUMMA) 112, Madrid
  - Hospital Universitario Quirón, Madrid

REFERENCES:
- [Background] Ibanez B, Prat-Gonzalez S, Speidl WS, Vilahur G, Pinero A, Cimmino G, Garcia MJ, Fuster V, Sanz J, Badimon JJ. Early metoprolol administration before coronary reperfusion results in increased myocardial salvage: analysis of ischemic myocardium at risk using cardiac magnetic resonance. Circulation. 2007 Jun 12;115(23):2909-16. doi: 10.1161/CIRCULATIONAHA.106.679639. Epub 2007 May 21. PMID 17515460
- [Background] Ibanez B, Cimmino G, Prat-Gonzalez S, Vilahur G, Hutter R, Garcia MJ, Fuster V, Sanz J, Badimon L, Badimon JJ. The cardioprotection granted by metoprolol is restricted to its administration prior to coronary reperfusion. Int J Cardiol. 2011 Mar 17;147(3):428-32. doi: 10.1016/j.ijcard.2009.09.551. Epub 2009 Nov 12. PMID 19913314
- [Background] Sharma SK, Kini A, Marmur JD, Fuster V. Cardioprotective effect of prior beta-blocker therapy in reducing creatine kinase-MB elevation after coronary intervention: benefit is extended to improvement in intermediate-term survival. Circulation. 2000 Jul 11;102(2):166-72. doi: 10.1161/01.cir.102.2.166. PMID 10889126
- [Background] Halkin A, Grines CL, Cox DA, Garcia E, Mehran R, Tcheng JE, Griffin JJ, Guagliumi G, Brodie B, Turco M, Rutherford BD, Aymong E, Lansky AJ, Stone GW. Impact of intravenous beta-blockade before primary angioplasty on survival in patients undergoing mechanical reperfusion therapy for acute myocardial infarction. J Am Coll Cardiol. 2004 May 19;43(10):1780-7. doi: 10.1016/j.jacc.2003.10.068. PMID 15145099
- [Background] Harjai KJ, Stone GW, Boura J, Grines L, Garcia E, Brodie B, Cox D, O'Neill WW, Grines C. Effects of prior beta-blocker therapy on clinical outcomes after primary coronary angioplasty for acute myocardial infarction. Am J Cardiol. 2003 Mar 15;91(6):655-60. doi: 10.1016/s0002-9149(02)03401-x. PMID 12633793
- [Background] Larose E, Rodes-Cabau J, Pibarot P, Rinfret S, Proulx G, Nguyen CM, Dery JP, Gleeton O, Roy L, Noel B, Barbeau G, Rouleau J, Boudreault JR, Amyot M, De Larochelliere R, Bertrand OF. Predicting late myocardial recovery and outcomes in the early hours of ST-segment elevation myocardial infarction traditional measures compared with microvascular obstruction, salvaged myocardium, and necrosis characteristics by cardiovascular magnetic resonance. J Am Coll Cardiol. 2010 Jun 1;55(22):2459-69. doi: 10.1016/j.jacc.2010.02.033. PMID 20510213
- [Background] Raman SV, Simonetti OP, Winner MW 3rd, Dickerson JA, He X, Mazzaferri EL Jr, Ambrosio G. Cardiac magnetic resonance with edema imaging identifies myocardium at risk and predicts worse outcome in patients with non-ST-segment elevation acute coronary syndrome. J Am Coll Cardiol. 2010 Jun 1;55(22):2480-8. doi: 10.1016/j.jacc.2010.01.047. PMID 20510215
- [Background] Ibanez B, Fuster V, Macaya C, Sanchez-Brunete V, Pizarro G, Lopez-Romero P, Mateos A, Jimenez-Borreguero J, Fernandez-Ortiz A, Sanz G, Fernandez-Friera L, Corral E, Barreiro MV, Ruiz-Mateos B, Goicolea J, Hernandez-Antolin R, Acebal C, Garcia-Rubira JC, Albarran A, Zamorano JL, Casado I, Valenciano J, Fernandez-Vazquez F, de la Torre JM, Perez de Prado A, Iglesias-Vazquez JA, Martinez-Tenorio P, Iniguez A. Study design for the "effect of METOprolol in CARDioproteCtioN during an acute myocardial InfarCtion" (METOCARD-CNIC): a randomized, controlled parallel-group, observer-blinded clinical trial of early pre-reperfusion metoprolol administration in ST-segment elevation myocardial infarction. Am Heart J. 2012 Oct;164(4):473-480.e5. doi: 10.1016/j.ahj.2012.07.020. PMID 23067904
- [Derived] Lorca R, Jimenez-Blanco M, Garcia-Ruiz JM, Pizarro G, Fernandez-Jimenez R, Garcia-Alvarez A, Fernandez-Friera L, Lobo-Gonzalez M, Fuster V, Rossello X, Ibanez B. Coexistence of transmural and lateral wavefront progression of myocardial infarction in the human heart. Rev Esp Cardiol (Engl Ed). 2021 Oct;74(10):870-877. doi: 10.1016/j.rec.2020.07.007. Epub 2020 Aug 24. English, Spanish. PMID 32855096
- [Derived] Podlesnikar T, Pizarro G, Fernandez-Jimenez R, Montero-Cabezas JM, Greif N, Sanchez-Gonzalez J, Bucciarelli-Ducci C, Marsan NA, Fras Z, Bax JJ, Fuster V, Ibanez B, Delgado V. Left ventricular functional recovery of infarcted and remote myocardium after ST-segment elevation myocardial infarction (METOCARD-CNIC randomized clinical trial substudy). J Cardiovasc Magn Reson. 2020 Jun 11;22(1):44. doi: 10.1186/s12968-020-00638-8. PMID 32522198
- [Derived] Podlesnikar T, Pizarro G, Fernandez-Jimenez R, Montero-Cabezas JM, Sanchez-Gonzalez J, Bucciarelli-Ducci C, Ajmone Marsan N, Fras Z, Bax JJ, Fuster V, Ibanez B, Delgado V. Effect of Early Metoprolol During ST-Segment Elevation Myocardial Infarction on Left Ventricular Strain: Feature-Tracking Cardiovascular Magnetic Resonance Substudy From the METOCARD-CNIC Trial. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 1):1188-1198. doi: 10.1016/j.jcmg.2018.07.019. Epub 2018 Sep 12. PMID 30219400
- [Derived] Sala-Vila A, Fernandez-Jimenez R, Pizarro G, Calvo C, Garcia-Ruiz JM, Fernandez-Friera L, Rodriguez MD, Escalera N, Palazuelos J, Macias A, Perez-Asenjo B, Fernandez-Ortiz A, Ros E, Fuster V, Ibanez B. Nutritional preconditioning by marine omega-3 fatty acids in patients with ST-segment elevation myocardial infarction: A METOCARD-CNIC trial substudy. Int J Cardiol. 2017 Feb 1;228:828-833. doi: 10.1016/j.ijcard.2016.11.214. Epub 2016 Nov 9. PMID 27888762
- [Derived] Mateos A, Garcia-Lunar I, Garcia-Ruiz JM, Pizarro G, Fernandez-Jimenez R, Huertas P, Garcia-Alvarez A, Fernandez-Friera L, Bravo J, Flores-Arias J, Barreiro MV, Chayan-Zas L, Corral E, Fuster V, Sanchez-Brunete V, Ibanez B; METOCARD-CNIC Investigators. Efficacy and safety of out-of-hospital intravenous metoprolol administration in anterior ST-segment elevation acute myocardial infarction: insights from the METOCARD-CNIC trial. Ann Emerg Med. 2015 Mar;65(3):318-24. doi: 10.1016/j.annemergmed.2014.07.010. Epub 2014 Aug 14. PMID 25129820
- [Derived] Pizarro G, Fernandez-Friera L, Fuster V, Fernandez-Jimenez R, Garcia-Ruiz JM, Garcia-Alvarez A, Mateos A, Barreiro MV, Escalera N, Rodriguez MD, de Miguel A, Garcia-Lunar I, Parra-Fuertes JJ, Sanchez-Gonzalez J, Pardillos L, Nieto B, Jimenez A, Abejon R, Bastante T, Martinez de Vega V, Cabrera JA, Lopez-Melgar B, Guzman G, Garcia-Prieto J, Mirelis JG, Zamorano JL, Albarran A, Goicolea J, Escaned J, Pocock S, Iniguez A, Fernandez-Ortiz A, Sanchez-Brunete V, Macaya C, Ibanez B. Long-term benefit of early pre-reperfusion metoprolol administration in patients with acute myocardial infarction: results from the METOCARD-CNIC trial (Effect of Metoprolol in Cardioprotection During an Acute Myocardial Infarction). J Am Coll Cardiol. 2014 Jun 10;63(22):2356-62. doi: 10.1016/j.jacc.2014.03.014. Epub 2014 Mar 30. PMID 24694530
- [Derived] Ibanez B, Macaya C, Sanchez-Brunete V, Pizarro G, Fernandez-Friera L, Mateos A, Fernandez-Ortiz A, Garcia-Ruiz JM, Garcia-Alvarez A, Iniguez A, Jimenez-Borreguero J, Lopez-Romero P, Fernandez-Jimenez R, Goicolea J, Ruiz-Mateos B, Bastante T, Arias M, Iglesias-Vazquez JA, Rodriguez MD, Escalera N, Acebal C, Cabrera JA, Valenciano J, Perez de Prado A, Fernandez-Campos MJ, Casado I, Garcia-Rubira JC, Garcia-Prieto J, Sanz-Rosa D, Cuellas C, Hernandez-Antolin R, Albarran A, Fernandez-Vazquez F, de la Torre-Hernandez JM, Pocock S, Sanz G, Fuster V. Effect of early metoprolol on infarct size in ST-segment-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention: the Effect of Metoprolol in Cardioprotection During an Acute Myocardial Infarction (METOCARD-CNIC) trial. Circulation. 2013 Oct 1;128(14):1495-503. doi: 10.1161/CIRCULATIONAHA.113.003653. Epub 2013 Sep 3. PMID 24002794
- See also: Related Info — http://www.cnic.es